CLINICAL TRIAL: NCT06179992
Title: A Cross-over Randomized-control Study Evaluating the Efficacy of GGED in Reducing Maladaptive Beliefs Related to Eating Disorders.
Brief Title: Study of the Efficacy of GGED: a Cognitive Training App for Eating Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María Roncero, Associate Professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GVA/2021/162
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-01

CONDITIONS: Eating Disorders
Keywords: maladaptive beliefs; cognitive therapy; mobile app; apps; e-health; non-clinical population
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: All participants were requested to complete web-based assessment, with questionnaires relating to maladaptive beliefs associated with ED, eating and emotional symptomatology, body satisfaction and self-esteem at baseline (T1). The experimental group started using the app for 15 days, and later completed the following assessment (T2). The control group also completed the T2 in the same date but started to use the app after this second assessment.15 days and one month later, both groups completed T3 and T4.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group used the GGED module for 15 days after the first assessment.
  Interventions: Device: GGED mobile app
- Control group (Active Comparator): The control group used the GGED module for 15 days after the second assessment.
  Interventions: Device: GGED mobile app

INTERVENTIONS:
Device: GGED mobile app — The intervention will be done through an app named GGED, which is used to work on the dysfunctional beliefs that are associated with eating disorders. The app is made up of a series of levels comprising the topics that are normally worked on in CBT in relation to eating disorders. At each level, affirmations in the form of beliefs appear on the screen, and the person must accept them if they are functional, adaptive and positive; or reject them if they are dysfunctional, maladaptive and negative.
  Other Names: GGED app

SUMMARY:
The aim of the present study is to evaluate the efficacy of GGTCA to decrease the maladaptive beliefs associated with eating disorders (ED) in non-clinical adult population. Specifically, a randomized controlled trial with crossover assignment design and two groups (experimental and control) will be carried out in adults aged 18-65 years to assess the changes pre and post use the app. It's expected that after the use of the GGTCA app for 15 days are, at the primary level: decrease in the degree of ascription to dysfunctional beliefs associated with ED; and at the secondary level: increase in self-esteem; decrease in eating symptomatology; and no changes in emotional symptomatology, since the pilot study did not find. These results are also expected to be maintained in subsequent follow-ups, at 15 days and a month after to finish the app in experimental group, and 15 days after to finish the app in control group.

DETAILED DESCRIPTION:
There is a digital platform called GGtude, which is composed of different modules, each of them aimed at working with different mental health problems. The goal is to provide an easy-to-use tool as a CBT complement to work on the self-dialogue that relates to the core beliefs associated with the psychological problem in particular. To achieve this target, a cognitive training exercise is performed: different sentences appear in the form of beliefs, and the person must identify and accept those beliefs that are functional, adaptive and positive, dragging them to the lower part of the screen; and reject those that are dysfunctional, maladaptive and negative dragging them to the upper part of the screen.

There are different modules, for example, to work self-esteem, depression, body image or obsessive-compulsive disorder, that have proven their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 40.
* Have a dispositive with Internet access.

Exclusion Criteria:

* None.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in the degree of ascription to dysfunctional beliefs associated with ED. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in the degree of ascription to dysfunctional beliefs associated with ED measured by the Eating Disorder Beliefs Questionnaire (EDBQ). It is composed of 32 items that examines core beliefs about weight, physical appearance and eating that are associated with eating disorders. Items are rated on an analog scale from 0 to 100, being 0 "I do not usually believe this at all" and 100 "I am usually completely convinced that this is true". Higher scores indicate the person has more degree of ascription to dysfunctional beliefs associated with eating disorders.
Change in maladaptive body and eating beliefs. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in maladaptive body and eating beliefs associated with ED measured by Obsessive Beliefs about Body Size and Eating Survey (OBBSES). It is composed of 57 items, which involve beliefs associated with food, eating, weight and body shape, divided into 5 factors: 1) appearance perfectionism; 2) vulnerability to weight gain; 3) eating control; 4) magical thinking; and, 5) thought control. People have to indicate in each item their degree of agreement in a Likert scale whit 7 point (1= "desagree very much" and 7 = "agree very much"). Higher scores indicate the person has more maladaptive body and eating beliefs.

SECONDARY OUTCOMES:
Change in eating symptomatology. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in eating symptoms measured by the Eating Disorder Examination Questionnaire (EDE-Q). It is a 36-item self-report questionnaire with 7-point Likert-type scale ranging from 0 (No day/ No time/ Not at all) to 6 (Every day/ Always/ Completely). It's composed of attitudinal and behavioral items, using for the present study only the attitudinal items (22 items). Higher scores indicate the person has greater presence of eating symptomatology.
Change in body satisfaction. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in body satisfaction measured by the Body Appreciation Scale-2 (BAS-2). It is a single-factor questionnaire that evaluates body satisfaction with 10 items on a 5-point Likert scale (1 = Never; 5 = Always). Higher scores indicate the person has more body satisfaction.
Change in self-esteem. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in self-report measures with The Single-Item Self-Esteem Scale (SISE; Robins et al., 2001). The person has to indicate how the statement "I have high self-esteem" describes him/her on a 9-point scale (1 = "Not very true for me" and 9 = "Very true for me"). Higher scores indicate the person has more self-esteem.
Change in emotional symptomatology. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in emotional symptomatology measured by The Depression, Anxiety-Stress Scale (DASS-21). It is composed of 21 items that evaluate emotional negative symptoms: depression, anxiety and stress. It has a Likert scale with 4 points (0 = "Did not apply to me at all" and 3 = "Applied to me very much or most of the time"). In this study only the scale of depression was used, composed of 7 items. Higher scores indicate the person has more emotional symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: 3 months after the study is published.
Access Criteria: The variables analyzed will be included in the manuscript in which the RCT data are presented, and will be published on the institutional page of the applicants' university (https://roderic.uv.es/) up to 3 months after the article is published.
URL: http://roderic.uv.es

REFERENCES:
- See also: Description Information about GGTUDE Mobile App and links to download. — http://ggapps.net/2018/04/11/ggro-relationship-obsession-rocd/

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT06179992/SAP_000.pdf
  • Informed Consent Form (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT06179992/ICF_001.pdf